CLINICAL TRIAL: NCT03641703
Title: An Open-Label, Multicentre, Long-Term Follow-Up Study to Investigate the Safety and Durability of Response Following Dosing of a Novel Adeno-Associated Viral Vector (FLT180a) in Patients With Haemophilia B
Brief Title: A Long-Term Follow-Up Study of Haemophilia B Patients Who Have Undergone Gene Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Freeline has decided to pause development of FLT180a for business priorities
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT180a-04
Record Dates: First submitted 2018-07-27; First posted 2018-08-22 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLT180a (Experimental): Participants who have received gene therapy vector (FLT180a)
  Interventions: Biological: FLT180a

INTERVENTIONS:
Biological: FLT180a — FLT180a is a replication-incompetent adeno-associated viral vector. The vector is composed of a DNA vector genome encapsidated in an adeno-associated virus derived protein capsid. The expression cassette contains DNA encoding Factor IX.

SUMMARY:
Severe haemophilia B (HB) is a bleeding disorder where a protein made by the body to help make blood clot is either partly or completely missing. This protein is called a clotting factor; with severe HB, levels of clotting Factor IX (nine; FIX) are very low and affected individuals can suffer life threatening bleeding episodes. HB mainly affects boys and men (approximately one in every 30,000 males). Current treatment for HB involves intravenous infusions of FIX as regular treatment (prophylaxis) or 'on demand' treatment. On demand treatment is highly effective at stopping bleeding but cannot fully reverse long-term damage that follows after a bleed. Regular treatment can prevent bleeding; however it is invasive for patients and also expensive.

This clinical study aims to investigate the long-term safety and durability of FIX activity in participants who have been dosed with a new gene therapy product (FLT180a) in earlier clinical studies. Following administration, FLT180a results in production of FIX in the participants' liver cells which is then released into the blood stream. The aim is to have the participants' own body produce levels of FIX that allow for clotting to occur as normal as would be seen in a non-HB individual. This would remove the need for prophylaxis or on demand treatment following just a single administration of FLT180a.

Up to 50 participants who have already been administered with FLT180a in the EU and US will take part in this study. Participants will be followed up in this trial until they have reached 15 years after being dosed. Participants will undergo procedures including physical examinations, join assessments, blood tests and liver ultrasounds. Participants will also need to complete a diary to document occurrence of bleeding episodes and record the amount of Factor IX concentrate they receive. Patient reports outcomes including measures of Quality of Life, disability and physical activity will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously received FLT180a within a clinical study.
* Able to give full informed consent and able to comply with all requirements of the study including long-term follow-up for the time frame the study requires.
* Willing to practice barrier contraception until at least three consecutive semen samples after vector administration are negative for vector sequences.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Primary Safety Measurement | From entry to 5 years post dosing
  Frequency of treatment-emergent adverse events/reactions (AE/ARs) reported according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or later (Primary Safety).
Durability of Response | From entry to 5 years post dosing
  Durability of response will be estimated by the rate of decline of the FIX activity observed from study entry (Primary Endpoint)

SECONDARY OUTCOMES:
Secondary Safety Measurement | From entry to 5 years post dosing
  Frequency of reporting of abnormal or change from baseline findings from safety assessments including laboratory assessments, vital signs, physical exam and liver ultrasound according to common terminology criteria for Adverse Events (CTCAE) version 5.0 or later.
FIX Activity Levels at or below 150% | From entry to 5 years post dosing
  Samples will be taken at each visit to measure FIX activity levels and the proportion of patients achieving FIX activity at or above 5%, 15%, 30%, 40%, 50%, 70% but no more than 150% of normal at each scheduled visit.
FIX Activity Levels including 150% or above | From entry to 5 years post dosing
  Samples will be taken at each visit to measure FIX activity levels and the proportion of patients achieving FIX activity at or above 5%, 15%, 30%, 40%, 50%, 70% and 150% of normal at each required visit.
FIX Activity Levels - Change from baseline | From entry to 5 years post dosing
  Change from baseline (prior to FLT180a dosing) in FIX activity at each scheduled visit.
Haemostatic Effectiveness - Bleeding Rates | From entry to 5 years post dosing
  Change from baseline (prior to FLT180a dosing) in annualised bleeding rate by measurement of number of breakthrough bleeding episodes.
Haemostatic Effectiveness - FIX Concentrate Consumption | From entry to 5 years post dosing
  Change from baseline (prior to FLT180a dosing) in FIX concentrate consumption by measurement of factor concentrate consumed by the patient.
FLT180a effectiveness related to surgical/dental procedures by assessment of consumption of exogenous clotting factors at Time of surgery, Time of drain removal (if applicable) | From entry to 5 years post dosing
  Consumption of exogenous clotting factors, related to an individual surgery, will be collected at the three time-points (time of surgery, time of drain removal (if applicable) and time of discharge or 6-days post surgery) for each surgery occurring from patient entry into trial until 5 years post-dosing.
FLT180a effectiveness related to surgical/dental procedures by assessment of measurement of absolute blood loss at Time of surgery, Time of drain removal (if applicable) | From entry to 5 years post dosing
  Measurement of absolute blood loss, related to an individual surgery, will be collected at the three time-points (Time of surgery, Time of drain removal (if applicable) and The earlier of discharge of 6-days post surgery) for each surgery occurring from patient entry into trial until 5 years post-dosing.
FLT180a effectiveness related to surgical/dental procedures by assessment of blood transfusion requirement, volume and number of transfusions at Time of surgery, Time of drain removal (if applicable) | From entry to 5 years post dosing
  Transfusion requirement (volume and number of transfusions), related to an individual surgery, will be collected at the three time-points (Time of surgery, Time of drain removal (if applicable) and The earlier of discharge of 6-days post surgery) for each surgery occurring from patient entry into trial until 5 years post-dosing.
FLT180a effectiveness related to surgical/dental procedures by assessment of efficacy of haemostasis as judged by surgeon on a 4-point scale at Time of surgery, Time of drain removal (if applicable) | From entry to 5 years post dosing
  Assessment of efficacy of haemostasis as judged by surgeon, related to an individual surgery, will be collected at the three time-points (Time of surgery, Time of drain removal (if applicable) and The earlier of discharge of 6-days post surgery) for each surgery occurring from patient entry into trial until 5 years post-dosing.
Immune response to the hFIX transgene product (i.e., development of inhibitors) will be assessed by measurement of the level of inhibitors. | From entry to 5 years post dosing
  Samples will be taken to capture development of inhibitors overtime.
Clearance of vector genomes (vgs) in plasma, urine, saliva, stool and semen. | From entry to complete clearance of vgs in all sample pools.
  Samples from each pool will be taken at each visit until there have been 3 consecutive samples that are negative for vgs.

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - The Haemophilia and Thrombosis Centre, Canterbury, Kent
  - Sheffield Teaching Hospital, Sheffield, South Yorkshire
  - Royal Free London NHS Foundation Tust, London
  - Newcastle Hemophilia Comprehensive Care Centre, Newcastle
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Southampton Haemophilia Comprehensive Care Centre, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chowdary P, Shapiro S, Makris M, Evans G, Boyce S, Talks K, Dolan G, Reiss U, Phillips M, Riddell A, Peralta MR, Quaye M, Patch DW, Tuddenham E, Dane A, Watissee M, Long A, Nathwani A. Phase 1-2 Trial of AAVS3 Gene Therapy in Patients with Hemophilia B. N Engl J Med. 2022 Jul 21;387(3):237-247. doi: 10.1056/NEJMoa2119913. PMID 35857660